CLINICAL TRIAL: NCT05215847
Title: A Phase 2 Open Label Study to Evaluate the Safety, Tolerability, and Efficacy of ARD-101 in Subjects At Least One Year After Bariatric Surgery
Brief Title: Study to Evaluate ARD-101 in Adults Receiving Bariatric Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aardvark Therapeutics, Inc. (Industry)
Collaborators: University of California, San Diego (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AARD-202
Record Dates: First submitted 2022-01-03; First posted 2022-01-31 (Actual); Results first posted 2024-11-14 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2024-10

CONDITIONS: Bariatric Surgery; Obesity; Weight Gain
Keywords: Obesity; Bariatric Surgery; Weight Gain; Anti-Obesity Agents
MeSH Terms: conditions — Obesity; Weight Gain

STUDY DESIGN:
Intervention Model Description: This study includes one intervention arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ARD-101 (Experimental): Dose 200 mg of ARD-101, twice daily for 28 days
  Interventions: Drug: ARD-101

INTERVENTIONS:
Drug: ARD-101 — Twice daily, oral administration

SUMMARY:
The purpose of this study is to evaluate safety and efficacy of twice-daily ARD-101 in subjects at least one year after bariatric surgery (sleeve gastrectomy or gastric bypass).

DETAILED DESCRIPTION:
This is a Phase 2, open-label study to investigate the safety and efficacy of twice-daily ARD-101 in subjects at least one year after bariatric surgery (sleeve gastrectomy or gastric bypass). This study has a planned enrollment of 30 subjects (approximately 15 for each preceding surgical procedure) and will be conducted in a single center in the United States.

The study will consist of a Screening Period (up to 28 days), a Treatment Period (28 days), and a Follow-up Period (EOS Visit within 14 days after receiving the last dose of ARD-101). The screening procedures will be initiated upon completion of the informed consent process. Following completion of screening procedures and confirmation of eligibility, subjects will be enrolled to receive ARD-101.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects, 18-75 years of age
* Willing and able to provide signed and dated informed consent prior to any study-related procedures and willing and able to comply with all study procedures
* Body Mass Index (BMI) of 35-60 kg/m2 during the Screening Period
* Status of at least 1-year post sleeve gastrectomy or gastric bypass surgery. Subjects must have a documented weight loss of at least 50% of their excess weight at their nadir, and must have regained at least 20% of their nadir weight loss. Excess weight is defined as maximum preoperative weight - weight corresponding to a BMI of 25 kg/m2
* Subjects with rescue surgery (e.g. gastric band to sleeve gastrectomy or gastric bypass; sleeve gastrectomy to gastric bypass) will be allowed, with time since second surgery of at least 12 months.
* Subjects with a history of revision procedures will be allowed if at least 6 months have passed since the procedure and weight has not deviated more than 5% in the 3 months prior to enrollment
* No abnormal findings or abnormalities of clinical significance in vital signs, physical examination, clinical laboratory tests (CBC, urinalysis, blood biochemistry, coagulation, pregnancy test (females), urine drug test, nicotine test, etc.), 12-lead electrocardiogram (ECG) during the Screening Period
* Serum creatinine, alkaline phosphatase, hepatic enzymes (aspartate aminotransferase, alanine aminotransferase) and total bilirubin (unless the subject has documented Gilbert syndrome) not exceeding 1.5-fold the upper laboratory norm and estimated Glomerular Filtration Rate (eGFR) >30 mL/min
* Standard 12-lead ECG parameters after 10minutes resting in supine position in the following ranges; 120 ms <PR <220 ms, QRS <120 ms, QTc <= 430 ms if male, <= 450 ms if female and normal ECG tracing unless the Investigator considers an ECG abnormality within described limits to be not clinically relevant
* Stable or well controlled blood pressure per Investigator's judgement during the Screening Period. Specifically: Vital signs after 10 minutes sitting in a chair (feet on floor, back supported):

  i. 95 mmHg < systolic blood pressure (SBP) <160 mmHg, ii. 45 mm Hg < diastolic blood pressure (DBP) <100 mm Hg, iii. 40 bpm < heart rate (HR) <100 bpm.
* Prediabetes- defined as a fasting blood glucose between 100-125 mg/dL OR an HbA1c between 5.7-6.5% at screening
* Type 2 diabetes- Defined as previous diagnosis by a healthcare professional OR a fasting blood glucose > 126 mg/dL OR HbA1c > 6.5% at screening.
* Patients with type 2 diabetes treated with metformin may be enrolled. However, patients with type 2 diabetes on any other therapy will be excluded.
* Female subjects must have negative serum pregnancy test and must not be lactating. For females able to bear children, a hormonal (i.e., oral, implantable, or injectable) and single barrier method (i.e., sponge), or a double-barrier method of birth control (i.e., condom with spermicide) or abstinence must be used/practiced throughout the study and for 90 days following last dose of study medication; for effective form of birth control.
* Females of non-childbearing potential, defined as surgically sterile (status post hysterectomy, bilateral oophorectomy, bilateral tubal ligation, bilateral salpingectomy, or bilateral tubal occlusion) or post-menopausal for at least 12 months (may be confirmed with a screening follicle stimulating hormone (FSH) level in the post-menopausal lab range), do not require contraception during the study.
* Males with female partners of childbearing potential must agree to a double-barrier method if participants become sexually active during the study and for 90 days following the last dose of the study medication. Male subjects must not donate sperm for 90 days following their participation in the study.

Exclusion Criteria:

* Any relevant gastrointestinal (GI) surgery (excluding the gastric bypass or sleeve gastrectomy) per Investigator judgement
* History of significant drug hypersensitivity or anaphylaxis
* Participation in a weight loss program or clinical trial for weight loss within the 3 months prior to enrollment
* Received any experimental drugs or devices or have participated in a clinical study within 30 days prior to enrollment
* Diabetes treatment (unless metformin as outlined), or chronic oral steroids, or treatment with immune modulators, anti-obesity drugs, chronic opiate therapy, or antipsychotic medications
* Currently receiving any drug-based therapy for weight management
* Thyroid-stimulating hormone (TSH) level is outside of normal limit during the Screening Period
* The presence of diseases with abnormal clinical manifestations that need to be excluded based on their possible contribution to weight loss or weight gain, including but not limited to nervous, cardiovascular, blood and lymphatic system, immune, renal, hepatic, gastrointestinal, respiratory, metabolic and skeletal diseases during the Screening Period
* History of myocardial infarction, unstable angina, arterial revascularization, stroke, New York Heart Association Functional Class II-IV heart failure, or transient ischemic attack within 6 months prior to Visit 1
* Any malignancy not considered cured (except focal, treated basal cell carcinoma and squamous cell carcinoma of the skin); a participant is considered cured if there has been no evidence of cancer recurrence in the previous 5 years
* History of major depressive disorder or history of other severe psychiatric disorders (e.g., schizophrenia or bipolar disorder) within the last 2 years.
* Donated ≥200 mL of blood (blood components) or had massive blood loss, received blood transfusion or blood products within 3 months prior to enrollment
* Planned sperm/egg donation within 6 months post enrollment
* Positive urine drug test (morphine, methamphetamine, ketamine, ecstasy, and cannabis) during the Screening Period
* History of consuming more than 14 units of alcoholic beverages per week or of alcoholism or drug/chemical/substance abuse within past 2 years prior to enrollment (Note: one unit = 12 ounces of beer, 4 ounces of wine or 1 ounce of spirits)
* Smoking any amount within 3 months prior to enrollment
* Excessive consumption of tea, coffee, and/or caffeinated beverages (more than 8 cups, 250 mL for each cup) every day within 3 months prior to enrollment
* Symptomatic viral, bacterial (including upper respiratory infection), or fungal (non-cutaneous) infection within 1 week prior to enrollment
* History of human immunodeficiency virus antibody, hepatitis C antibody or hepatitis B virus surface antigen
* A history of psychiatric and psychological condition that, in the judgment of the investigator, may interfere with the planned treatment and follow-up, affect subject compliance or place the subject at high risk from treatment-related complications
* Poor venous access or inability to tolerate venipuncture
* Any condition or active drug treatment that the investigator or primary physician believes may not be appropriate for participating in the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-02-03 (Actual); Study Completion 2023-02-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Altman Clinical and Translational Research Institute, University of California, San Diego, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ARD-101
Started | 12
Completed | 11
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Population: Patients who completed treatment of ARD-101
Arm/Group | ARD-101
Number analyzed (Participants) | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 41 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 9
  More than one race | 0
  Unknown or Not Reported | 1
Weight [Mean (Standard Deviation); unit: Kilograms] | 117.9 (21.8)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 42.7 (4.98)
Height [Mean (Standard Deviation); unit: Centimeter] | 165.6 (9.7)

OUTCOME MEASURES:

1. Primary Outcome: Relative Change in Body Weight (%)
Description: The percent total weight change at the end of treatment from baseline
Time Frame: Baseline and Day 28
Population: Participants that have completed dosing with ARD-101.
Measure: Mean (Standard Deviation); unit: Percent Change
Groups:
- ARD-101: ARD-101 200 mg, orally twice daily for 28 days
Arm/Group | ARD-101
Number analyzed (Participants) | 11
Percent Change | 0.033 (1.515)

2. Secondary Outcome: Incidence of Treatment-emergent Adverse Events (TEAE)
Description: The incidence of treatment-emergent adverse events (TEAE) during the treatment period
Time Frame: Days 1-28
Population: Safety analysis set. All participants that have been dosed with ARD-101.
Measure: Count of Participants; unit: Participants
Arm/Group | ARD-101
Number analyzed (Participants) | 12
Participants | 6
Statistical Analysis 1: Comparison: ARD-101; Test type: Other — Adverse event subject incidence and event frequency; Adverse event subject incidence and event frequency

3. Secondary Outcome: Change in Blood Lipid Concentrations
Description: The change in blood lipid concentrations (total cholesterol, triglyceride, high density lipoprotein cholesterol, and low-density lipoprotein cholesterol) at the end of treatment from the baseline
Time Frame: Run-in Visit (baseline), Day 28
Population: All subjects who completed dosing of ARD-101.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | ARD-101
Number analyzed (Participants) | 11
mg/dL
  Total Cholesterol | -0.73 (18.23)
  Triglyceride | 2.09 (32.14)
  High density lipoprotein cholesterol | -0.82 (9.36)
  Low-density lipoprotein cholesterol | -0.36 (15.58)

4. Secondary Outcome: Change in Waist Circumference
Description: The change in waist circumference from baseline to end of treatment
Time Frame: Baseline and Day 28
Population: One participant was removed from waist circumference analysis due to improper measurement documentation by the study site.
Measure: Mean (Standard Deviation); unit: Centimeters
Arm/Group | ARD-101
Number analyzed (Participants) | 10
Centimeters | -0.7 (1.03)

5. Secondary Outcome: Change in Hemoglobin A1c
Description: The change in glycated hemoglobin (HbA1c) at the end of treatment from the baseline
Time Frame: Screening (baseline), Day 28
Population: One subject did not have their HbA1c collected/documented, so no data was provided to include in analysis.
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | ARD-101
Number analyzed (Participants) | 10
Percentage | 0.04 (0.17)

6. Other Pre Specified Outcome: Categorical Weight Loss
Description: Proportion of subjects who lose < 5% and ≥ 5% initial weight
Time Frame: Run-in Visit (baseline), Day 28
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Circulating Levels of Glucagon-like Peptide (GLP)-1 (Pmol) During Mixed-Meal Tolerance Test (MMTT) at Baseline and on Day 28, and Prior to and Post Dosing on Day 1
Description: Circulating levels of glucagon-like peptide (GLP)-1 (pmol) prior to (negative timepoints) and post (positive timepoints) the Ensure meal given for mixed-meal tolerance test (MMTT) at baseline (run-in visit) and on day 28, and pre-dosing and 1 and 2 hours post the first dosing on day 1.
Time Frame: Run-in Visit (baseline), Day 1, Day 28
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Circulating Levels of Cholecystokinin (CCK) (pg/mL) During MMTT at Baseline and on Day 28, and Prior to and Post Dosing on Day 1
Description: Circulating levels of cholecystokinin (CCK) (pg/mL) prior to (negative timepoints) and post (positive timepoints) the Ensure meal given for MMTT at baseline (run-in visit) and on day 28, and pre-dosing and 1 and 2 hours post the first dosing on day 1.
Time Frame: Run-in Visit (baseline), Day 1, Day 28
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Circulating Levels of Peptide YY (PYY) (pg/mL) During MMTT at Baseline and on Day 28, and Prior to and Post Dosing on Day 1
Description: Circulating levels of peptide YY (PYY) (pg/mL) prior to (negative timepoints) and post (positive timepoints) the Ensure meal given for MMTT at baseline (run-in visit) and on day 28, and pre-dosing and 1 and 2 hours post the first dosing on day 1.
Time Frame: Run-in Visit (baseline), Day 1, Day 28
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Circulating Levels of Amylin (Pmol) During MMTT at Baseline and on Day 28, and Prior to and Post Dosing on Day 1
Description: Circulating levels of amylin (pmol) prior to (negative timepoints) and post (positive timepoints) the Ensure meal given for MMTT at baseline (run-in visit) and on day 28, and pre-dosing and 1 and 2 hours post the first dosing on day 1.
Time Frame: Run-in Visit (baseline), Day 1, Day 28
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Circulating Levels of Glucose-dependent Insulinotropic Polypeptide (GIP) (pg/mL) During MMTT at Baseline and on Day 28, and Prior to and Post Dosing on Day 1
Description: Circulating levels of glucose-dependent insulinotropic polypeptide (GIP) (pg/mL) prior to (negative timepoints) and post (positive timepoints) the Ensure meal given for MMTT at baseline (run-in visit) and on day 28, and pre-dosing and 1 and 2 hours post the first dosing on day 1.
Time Frame: Run-in Visit (baseline), Day 1, Day 28
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Circulating Levels of Ghrelin (pg/mL) During MMTT at Baseline and on Day 28, and Prior to and Post Dosing on Day 1
Description: Circulating levels of ghrelin (pg/mL) prior to (negative timepoints) and post (positive timepoints) the Ensure meal given for MMTT at baseline (run-in visit) and on day 28, and pre-dosing and 1 and 2 hours post the first dosing on day 1.
Time Frame: Run-in Visit (baseline), Day 1, Day 28
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Circulating Levels of Leptin (ng/mL) During MMTT at Baseline and on Day 28, and Prior to and Post Dosing on Day 1
Description: Circulating levels of leptin (ng/mL) prior to (negative timepoints) and post (positive timepoints) the Ensure meal given for MMTT at baseline (run-in visit) and on day 28, and pre-dosing and 1 and 2 hours post the first dosing on day 1.
Time Frame: Run-in Visit (baseline), Day 1, Day 28
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Circulating Levels of Adiponectin (mcg/mL) During MMTT at Baseline and on Day 28, and Prior to and Post Dosing on Day 1
Description: Circulating levels of adiponectin (mcg/mL) prior to (negative timepoints) and post (positive timepoints) the Ensure meal given for MMTT at baseline (run-in visit) and on day 28, and pre-dosing and 1 and 2 hours post the first dosing on day 1.
Time Frame: Run-in Visit (baseline), Day 1, Day 28
Reporting Status: Not Posted

15. Other Pre Specified Outcome: Circulating Levels of Glucagon (pg/mL) During MMTT at Baseline and on Day 28, and Prior to and Post Dosing on Day 1
Description: Circulating levels of glucagon (pg/mL) prior to (negative timepoints) and post (positive timepoints) the Ensure meal given for MMTT at baseline (run-in visit) and on day 28, and pre-dosing and 1 and 2 hours post the first dosing on day 1.
Time Frame: Run-in Visit (baseline), Day 1, Day 28
Reporting Status: Not Posted

16. Other Pre Specified Outcome: Serum Levels of Glucose (mg/dL) During MMTT at Baseline and on Day 28
Description: Serum levels of glucose (mg/dL) prior to (negative timepoints) and post (positive timepoints) the Ensure meal given for MMTT at baseline (run-in visit) and on day 28.
Time Frame: Run-in Visit (baseline), Day 28
Reporting Status: Not Posted

17. Other Pre Specified Outcome: Serum Levels of Insulin (uIU/mL) During MMTT at Baseline and on Day 28
Description: Serum levels of insulin (uIU/mL) prior to (negative timepoints) and post (positive timepoints) the Ensure meal given for MMTT at baseline (run-in visit) and on day 28.
Time Frame: Run-in Visit (baseline), Day 28
Reporting Status: Not Posted

18. Other Pre Specified Outcome: Serum Levels of C-peptide (ng/mL) During MMTT at Baseline and on Day 28
Description: Serum levels of C-peptide (ng/mL) prior to (negative timepoints) and post (positive timepoints) the Ensure meal given for MMTT at baseline (run-in visit) and on day 28.
Time Frame: Run-in Visit (baseline), Day 28
Reporting Status: Not Posted

19. Other Pre Specified Outcome: Serum Levels of Free Fatty Acids During MMTT at Baseline and on Day 28
Description: Serum levels of free fatty acids (FFA) prior to (negative timepoints) and post (positive timepoints) the Ensure meal given for MMTT at baseline (run-in visit) and on day 28.
Time Frame: Run-in Visit (baseline), Day 28
Reporting Status: Not Posted

20. Other Pre Specified Outcome: Circulating Levels of Interleukin (IL)-1 Beta (pg/mL) During MMTT
Description: Circulating levels of interleukin (IL)-1 beta (pg/mL) at run in visit and end of treatment (day 28) performed during the MMTT
Time Frame: Run-in Visit (baseline), Day 28
Reporting Status: Not Posted

21. Other Pre Specified Outcome: Circulating Levels of IL-6 (pg/mL) During MMTT
Description: Circulating levels of IL-6 (pg/mL) at run in visit and end of treatment (day 28) performed during the MMTT
Time Frame: Run-in Visit (baseline), Day 28
Reporting Status: Not Posted

22. Other Pre Specified Outcome: Circulating Levels of IL-10 (pg/mL) During MMTT
Description: Circulating levels of IL-10 (pg/mL) at run in visit and end of treatment (day 28) performed during the MMTT
Time Frame: Run-in Visit (baseline), Day 28
Reporting Status: Not Posted

23. Other Pre Specified Outcome: Circulating Levels of IL-12 p40 (pg/mL) During MMTT
Description: Circulating levels of IL-12 p40 (pg/mL) at run in visit and end of treatment (day 28) performed during the MMTT
Time Frame: Run-in Visit (baseline), Day 28
Reporting Status: Not Posted

24. Other Pre Specified Outcome: Circulating Levels of IL-12 p70 (pg/mL) During MMTT
Description: Circulating levels of IL-12 p70 (pg/mL) at run in visit and end of treatment (day 28) performed during the MMTT
Time Frame: Run-in Visit (baseline), Day 28
Reporting Status: Not Posted

25. Other Pre Specified Outcome: Circulating Levels of IL-17 (pg/mL) During MMTT
Description: Circulating levels of IL-17 (pg/mL) at run in visit and end of treatment (day 28) performed during the MMTT
Time Frame: Run-in Visit (baseline), Day 28
Reporting Status: Not Posted

26. Other Pre Specified Outcome: Circulating Levels of Tumor Necrosis Factor (TNF)-Alpha (pg/mL) During MMTT
Description: Circulating levels of tumor necrosis factor (TNF)-alpha (pg/mL) at run in visit and end of treatment (day 28) performed during the MMTT
Time Frame: Run-in Visit (baseline), Day 28
Reporting Status: Not Posted

27. Other Pre Specified Outcome: Circulating Levels of C Reactive Protein (CRP) (mg/L) During MMTT
Description: Circulating levels of C reactive protein (CRP) (mg/L) at run in visit and end of treatment (day 28) performed during the MMTT
Time Frame: Run-in Visit (baseline), Day 28
Reporting Status: Not Posted

28. Other Pre Specified Outcome: Body Fat Percentage
Description: Body fat percentage measured by bioelectrical impedance scale
Time Frame: Run-in Visit (baseline), Days 1-28
Reporting Status: Not Posted

29. Other Pre Specified Outcome: Change in the Percentage of Liver Fat Content
Description: Change in the percentage of liver fat content assessed by magnetic resonance imaging-derived proton density fat fraction (MRI-PDFF)
Time Frame: Run-in Visit (baseline), Day 28
Reporting Status: Not Posted

30. Other Pre Specified Outcome: Change in Homeostatic Model Assessment for Insulin Resistance (HOMA-IR)
Description: The change in homeostatic model assessment for insulin resistance (HOMA-IR) at the end of treatment from the baseline
Time Frame: Run-in Visit (baseline), Day 28
Reporting Status: Not Posted

31. Other Pre Specified Outcome: Change in Fasting Blood Glucose
Description: The change in fasting blood glucose at the end of treatment from the baseline
Time Frame: Run-in Visit (baseline), Day 28
Reporting Status: Not Posted

32. Other Pre Specified Outcome: Change in Serum Bile Acids
Description: Change in serum bile acids at the end of treatment compared to the baseline
Time Frame: Run-in Visit (baseline), Day 28
Reporting Status: Not Posted

33. Other Pre Specified Outcome: Phenotypic Taste Test
Description: Phenotypic taste test (using commercially available test strips) at baseline
Time Frame: Run-in Visit (baseline)
Reporting Status: Not Posted

34. Other Pre Specified Outcome: Control of Eating and Food Cravings
Description: Control of eating and food craving assessed by the Control of Eating Questionnaire (CoEQ), which is a 21-item questionnaire designed to assess the intensity and type of food cravings and subjective sensations of appetite and mood according to an individual's experience over the last 7 days. Items on the CoEQ are assessed by 100-mm visual analogue scales (VAS). Subjects will mark their level with a vertical line on the horizontal line of the VAS scale. The numerical value will start at 1.0 cm and end 10.0 cm. Use a ruler to determine the numerical value (to the tenth decimal) associated with the line marked by subjects. Higher score indicates less control of eating and food cravings.
Time Frame: Screening, Days 1, 15, and 28
Reporting Status: Not Posted

35. Other Pre Specified Outcome: Change in Indirect Calorimetry
Description: Change in indirect calorimetry between Day 1 and Day 28
Time Frame: Day 1, Day 28
Reporting Status: Not Posted

36. Other Pre Specified Outcome: Area Under the Curve (AUC) of Serum Level of Glucose (mg/dL) During MMTT
Description: Changes in AUC of serum level of glucose (mg/dL) during MMTT between baseline and Day 28
Time Frame: Run-in Visit (baseline), Day 28
Reporting Status: Not Posted

37. Other Pre Specified Outcome: Area Under the Curve (AUC) of Serum Level of Insulin (uIU/mL) During MMTT
Description: Changes in AUC of serum level of insulin (uIU/mL) during MMTT between baseline and Day 28
Time Frame: Run-in Visit (baseline), Day 28
Reporting Status: Not Posted

38. Other Pre Specified Outcome: Area Under the Curve (AUC) of Serum Level of C-peptide (ng/mL) During MMTT
Description: Changes in AUC of serum levels of C-peptide (ng/mL) during MMTT between baseline and Day 28
Time Frame: Run-in Visit (baseline), Day 28
Reporting Status: Not Posted

39. Other Pre Specified Outcome: Changes in Fecal Microbial Species and Their Relative Abundance
Description: Changes in fecal microbial species and their relative abundance assessed by 16S rRNA gene sequencing
Time Frame: Day 1, Day 28
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: Any untoward event occurring in the clinical study framework was documented and recorded as an adverse event, including those occurring during treatment-free periods (including screening or post-treatment follow-up periods). Adverse event monitoring was performed and collected at screening, Day 1 (predose), Day 15, Day 28, and follow-up/end of study.
Arm/Group | ARD-101
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 6/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ARD-101 (N=12)
Mild Nausea (Gastrointestinal disorders) | 2 (2) — Related, no action was taken, resolved without sequelae
Mild Emesis (Gastrointestinal disorders) | 1 (1) — Related, no action was taken, resolved without sequelae
Mild Common Cold (Infections and infestations) | 1 (1) — No related, concomitant therapy intervention, resolved without sequelae
Mild Headache (Nervous system disorders) | 1 (2) — Related, no action was taken, resolved without sequelae
Mild Constipation (Gastrointestinal disorders) | 1 (1) — Related, no action was taken, resolved without sequelae
Mild Heart Burn (Gastrointestinal disorders) | 1 (1) — Related, no action was taken, resolved without sequelae
Mild Hypoglycemia (Endocrine disorders) | 1 (1) — Not related, no action was taken, resolved without sequelae
Mild COVID-19 (Infections and infestations) | 1 (1) — Not related, concomitant therapy intervention, resolved without sequelae
Mild Dyspepsia (Gastrointestinal disorders) | 1 (1) — Related, no action was taken, resolved without sequelae

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-09): https://cdn.clinicaltrials.gov/large-docs/47/NCT05215847/Prot_SAP_000.pdf